CLINICAL TRIAL: NCT06641479
Title: JiAngSu Maternal and INfant HEalth Database(JASMINE): Using Electronic Health Records to Improve Maternal and Child Health Care and Outcomes in China
Brief Title: JiAngSu Maternal and INfant HEalth Database
Acronym: JASMINE
Status: Active, not recruiting | Type: Observational
Sponsor: Yang Zhao (Other)
Collaborators: Ningbo University (Other)
Responsible Party: Sponsor-Investigator, Yang Zhao, Professor, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Other Study IDs: NMU-2024-808
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pregnant Women; Children
Keywords: Population-based healthcare database; Longitudinal study; Ambispective Cohort; Pregnant women and offspring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women and their offspring

SUMMARY:
With the implementation of China's universal two-child policy and a notable rise in adverse pregnancy outcomes, leveraging electronic health records (EHR) has become crucial for enhancing maternal health. Given the mature construction of the information platform and the well-established maternal and child health service system in Jiangsu Province, this study used the Jiangsu Health Information Platform to carry out the research on the JiAngSu Maternal and INfant hEalth database (JASMINE), which involved over 1.5 million mother-child pairs in Jiangsu Province.

JASMINE enables longitudinal follow-up of pregnant women and their offspring, facilitating the exploration of early-life exposures and their long-term outcomes through comprehensive data linkage. This longitudinal approach helps to clarify the relationship and etiological significance of risk factors associated with adverse pregnancy outcomes.It also permits the exploration of the health trajectory of women and children throughout their lives.

From January 2020 to December 2023, JASMINE has recorded extensive maternal and child health data, including socio-demographics, healthcare services, medications, and clinical outcomes.Additionally, it contains longitudinal measurements on risk factors for adverse pregnancy outcomes, which provides a robust foundation for future real-world studies of dynamic predictive models. This study has been approved approved by the Institutional Review Board of Nanjing Medical University.

Ultimately, this research aims to identify key predictors of adverse pregnancy outcomes and inform public health policies to improve maternal and child health in Jiangsu Province. Future directions will include developing targeted interventions based on study findings to enhance health outcomes for mothers and infants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and their offspring who registered at the Jiangsu maternal and child health information platform.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All pregnant women and their offspring registered at the Jiangsu maternal and child health information platform were enrolled.
Study Population: Pregnant women and their offspring who registered at the Jiangsu maternal and child health information platform.
Sampling Method: Non-Probability Sample
Enrollment: 1570360 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of preterm birth | Up to 42 weeks
  Regular contractions accompanied by cervical change at less than 37 weeks' gestation.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O60.
Incidence of pre-eclampsia | Up to 42 weeks
  New onset hypertension (>140 mm Hg systolic or >90 mm Hg diastolic) after 20 weeks of pregnancy and the coexistence of one or both of the following new-onset conditions: proteinuria (urine protein:creatinine ratio ≥30 mg/mmol, or albumin: creatinine ratio ≥8 mg/mmol, or ≥1 g/L [2+] on dipstick testing), other maternal organ dysfunction, including features such as renal or liver involvement, neurological or haematological complications, or uteroplacental dysfunction (such as fetal growth restriction, abnormal umbilical artery Doppler waveform analysis, or stillbirth).
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O14.
Incidence of eclampsia | Up to 42 weeks
  The occurrence of new-onset, generalized, tonic-clonic seizures or coma in a patient with preeclampsia or gestational hypertension.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O15.
Incidence of gestational diabetes mellitus | Up to 42 weeks
  Impaired Glucose Tolerance (IGT) with onset or first recognition during pregnancy.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O24.4.
Incidence of low birth weight | Up to 42 weeks
  Weight at birth of < 2500 g. Or, at least one of the following diagnoses in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : P07.0, P07.1.
Incidence of small for gestational age | Up to 42 weeks
  Less than the tenth birth weight centile using INTERGROWTH-21st. Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : P05.
Incidence of autism | Up to 10 years
  The following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : F84.
Incidence of birth defects | Up to 10 years
  Birth defects such as congenital malformations of the nervous system, congenital malformations of eye, ear, face and neck, congenital malformations of the circulatory system, congenital malformations of the respiratory system, or other birth defects.
  Or, at least one of the following diagnoses in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : Q00-Q99.
Incidence of postpartum hemorrhage | Within 24 hours after delivery
  Blood loss exceeding 500 mL following vaginal birth and 1000 mL following cesarean.
  Or, the following diagnose in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O72.
Incidence of stillbirth | Up to 42 weeks
  Death of a fetus that has reached a birth weight of 500 g, or if birth weight is unavailable, gestational age of 22 weeks or crown-to-heel length of 25 cm.
  Or, at least one of the following diagnoses in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : Z37.1, Z37.3, Z37.4, Z37.7.
Incidence of ruptured uterus | Up to 42 weeks
  Uterine rupture is confirmed by laparotomy. Or, at least one of the following diagnoses in the electronic health records according to the International Classification of Diseases 10th Revision (ICD-10) : O71.0, O71.1, O34.5, O62.4.
Incidence of maternal death | Up to 52 weeks
  Death of women while pregnant or within 42 days of termination of pregnancy irrespective of the site and size of pregnancy but related to or aggravated by the pregnancy or its management but not from accidental or incidental causes.
Incidence of neonatal death | Within 28 days after delivery
  Deaths among live births during the first 28 completed days of life

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Medical University, Nanjing, Jiangsu, China